CLINICAL TRIAL: NCT03113292
Title: Effectiveness and Cost-effectiveness of the Pilates Method Versus Home-based Exercises in Individuals With Chronic Non-specific Low Back Pain: a Randomized Controlled Trial
Brief Title: Effects of the Pilates Method Versus Home Exercise in Individuals With Chronic Non-specific Back Pain
Acronym: COmEBACK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Brasilia (Other)
Responsible Party: Principal Investigator, Prof. Rodrigo Luiz Carregaro, Prof. Dr., University of Brasilia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COmEBACK Trial; CAAE68870317.0.0000.8093 (Other: Ethics Commitee FCE/UnB)
Record Dates: First submitted 2017-04-02; First posted 2017-04-13 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Chronic Low Back Pain
Keywords: physical therapy; therapeutic exercises; low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Exercise Movement Techniques; Exercise Therapy

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled clinical trial, characterized by the application of therapeutic exercises, in which subjects will be randomly allocated into two groups: Pilates Method and Home-Based Exercises. The participantes will be individuals with non-specific chronic low back pain. The study will be reported following the recommendations of the CONSORT Statement. For the present study, chronic non-specific back pain was defined as uninterrupted low back pain for more than 12 weeks, with unknown causes.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor won't have any knowledge about the study purposes and will be unaware of the group allocation. The statistical analysis will also be performed blinded for group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates Method (Experimental): Mat Pilates Program, 2x/week, for 6 weeks, supervised by a Physiotherapist. Sessions will last forty five min, with 4 individuals per session. On average, 10 to 15 exercises will be performed per session, with repetitions ranging from 10 to 20 times, according subject's limitations. If necessary, the exercises will be adapted individually for the three levels of difficulty: basic, intermediate and advanced. Progress will be dependent on the absence of postural compensations when performing the repetitions of the exercises.
  Interventions: Other: Pilates
- Home Exercise Prescription (Active Comparator): Composed by two familiarization sessions, supervised by a Physiotherapist. The protocol include postural reeducation exercises, stretching and muscle strengthening, stabilization and mobilization of the spine. Subsequently, participants will receive an educational booklet containing information on low back pain, anatomy of the spine and its relation to the muscular chain, care during daily life activities and the importance of regular physical exercises. Also, it will include a booklet with the prescription of therapeutic home exercises to be performed during the next 6 weeks. It will be recommended that the participants perform the exercises 2x/week. Participants will also be contacted weekly by email and/or telephone, for remote supervision and for checking the prescribed exercises.
  Interventions: Other: Home Exercises

INTERVENTIONS:
Other: Pilates — The protocol will be composed by the following exercises, structured in each session according to progression, difficulty and focus (respiration, stability, muscle strength and joint mobility): Arm Arcs, Bent Knee Opening, Sidelying, Dead Bug, Femur Arcs, Quadruped Series, Single Leg Stretch, Prone Press Up, Sidekick (Front to Back 1 e 2), Leg Pull Front, Mermaid, Spine Stretch, The Hundred, Pelvic Clock, Bridging, Stanging Roll Down, Swan, Saw, Dart, Swimming, Book Opening.
  .
  Other Names: Therapeutic exercise
  Arms: Pilates Method
Other: Home Exercises — The protocol will be divided into 3 phases, each one composed by the following exercises and structured according to difficulty progression and focus (postural reeducation, muscle strength, balance, joint flexibility): Muscle strength exercises composed by abdominal exercises; back extension exercises; gluteus maximus exercises. Stretching exercises for the lower back, pelvis, iliopsoas muscle, tensor fascia latae muscle).
  Other Names: Therapeutic exercise
  Arms: Home Exercise Prescription

SUMMARY:
The aim is to compare the effectiveness and cost-effectiveness of a Pilates program versus home-based exercises in individuals with chronic non-specific low back pain. This is a randomized controlled trial with economic evaluation. Participants will be sequentially enrolled and randomly allocated into two groups: 1) Pilates: Mat Pilates sessions, supervised by a physiotherapist (2x/week for 6 weeks); 2) Home-Based Exercise: face-to-face familiarization (two sessions), supervised by another physiotherapist. After familiarization, the exercises will be prescribed using a booklet containing descriptions of sets/repetitions, as well as guidelines and precautions, to be performed during 6 weeks (2x/week) and monitored in a diary. Participants will be supervised by the physiotherapist (telephone/text messaging). Participants will be evaluated in three different moments: 1) Baseline (pre-intervention); 2) At the end of the intervention (post-intervention, 6 weeks); and 3) After six months follow-up (from post-intervention). Primary outcomes: pain intensity and disability. Secondary outcomes: perception of recovery, postural balance, and quality of life. Concurrently, a cost-effectiveness study will be conducted comparing the Pilates vs Home-Based Exercise, from the perspectives of public healthcare and society. In the first perspective, only costs incurred by the public healthcare system will be included (direct costs related to consultations, medications, tests, hospitalizations, and professional fees). In the second perspective, private health care expenses, costs incurred by patients (transportation and support by caregivers, when applicable), as well as indirect costs (missed workdays and loss of productivity) will be included. The incremental cost-effectiveness ratios for the primary outcomes and cost-utility ratios will be calculated for both perspectives. The cost-utility ratio will express the incremental costs per quality-adjusted life year (QALY). In addition, the absolute and incremental net monetary benefit will be calculated. Sensitivity analyses will be conducted. Data normality assumptions will be evaluated using the Shapiro Wilk test. If confirmed, a mixed model will be used, for the comparisons between groups and moments. It is hypothesized that the Pilates will be more cost-effective compared to the home-based exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Presence of chronic non-specific back pain for more than 12 consecutive weeks;
* Not having attended Pilates or physiotherapy sessions for at least 6 months prior to enrollment.

Exclusion Criteria:

* History of trauma or fractures in the spine;;
* Diagnosis of osteoarthritis, disc herniation or spondylolisthesis;
* Referred pain (visceral, abdominoplasty, appendicitis, abdominal and pelvic surgeries);
* Previous surgery on the spine;
* Presence of root symptoms;
* Pregnancy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 145 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Pain Intensiy | Change from Pre-Intervention (baseline) compared to Post-Intervention (6 weeks) and Follow-up (6 months)
  Pain Intensity measured on a Visual Analog Scale (VAS, in centimeters)
Disability | Change from Pre-Intervention (baseline) compared to Post-Intervention (6 weeks) and Follow-up (6 months)
  Quebec Back Pain Disability Scale, scores ranging from 0 to 100

SECONDARY OUTCOMES:
Health status | Change from Pre-Intervention (baseline) compared to Post-Intervention (6 weeks) and Follow-up (6 months)
  Measure of health status by the EQ-5D-3L questionnaire, consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which can take one of five responses. The responses record five levels of severity (no problems/slight problems/moderate problems/severe problems/extreme problems).
Balance | Change from Pre-Intervention (baseline) compared to Post-Intervention (6 weeks) and Follow-up (6 months)
  Balance Platform, variation of the platform displacement
Perception of Recovery | Change from Pre-Intervention (baseline) compared to Post-Intervention (6 weeks) and Follow-up (6 months)
  Perception of Recovery measured by a Global Perceived Effect Scale (11-point scale), ranging from -5 ("much worse"), 0 ("no change"), to 5 ("completely recovered")

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo L Carregaro, PhD, Principal Investigator — University of Brasilia, School of Physical Therapy
Locations (1):
- Campus UnB Ceilândia, Brasília, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boff TA, Pasinato F, Ben AJ, Bosmans JE, van Tulder M, Carregaro RL. Effectiveness of spinal manipulation and myofascial release compared with spinal manipulation alone on health-related outcomes in individuals with non-specific low back pain: randomized controlled trial. Physiotherapy. 2020 Jun;107:71-80. doi: 10.1016/j.physio.2019.11.002. Epub 2019 Nov 18. PMID 32026838